CLINICAL TRIAL: NCT04521738
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Subcutaneous Doses of SAR441255 in Lean to Overweight Adult Subjects
Brief Title: First-in-human Study to Assess Safety and Tolerability of a Single Subcutaneous Dose of SAR441255 in Lean to Overweight Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TDU15478; U1111-1210-0180 (Other: UTN)
Record Dates: First submitted 2020-08-19; First posted 2020-08-20 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Overweight; Healthy Subjects
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR441255 (Experimental): Single dose, subcutaneous, escalating dose
  Interventions: Drug: SAR441255
- Placebo (Placebo Comparator): Single dose, subcutaneous, matched volume
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SAR441255 — Pharmaceutical form:solution for injection
  Route of administration: subcutaneous
  Arms: SAR441255
Drug: placebo — Pharmaceutical form:solution for injection
  Route of administration: subcutaneous
  Arms: Placebo

SUMMARY:
Primary Objective:

To assess the safety and tolerability of SAR441255 after ascending single subcutaneous (SC) doses

Secondary Objectives:

To assess the pharmacokinetic parameters of SAR441255 in plasma after ascending single SC doses

To assess the pharmacodynamic effects on glycemic parameters (fasting and postprandial glucose, C-peptide and insulin)

DETAILED DESCRIPTION:
Study duration per participant is approximately 8 weeks including a 21-day screening and baseline phase, a 4-day treatment phase and a 28-day follow up period after dosing.

ELIGIBILITY:
Inclusion criteria :

* Male and female subjects, between 18 and 55 years of age, inclusive
* Body Mass Index ≥20 and ≤30 kg/m2
* Body weight between 65 and 90 kg, inclusive
* No concomitant medication
* Fasting Plasma Glucose <126 mg/dL
* Hemoglobin A1c <6.5%
* Triglycerides <300 mg/dL
* Low-density lipoprotein (LDL) Cholesterol <200 mg/dL
* Permanent sterile or postmenopausal, if female

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, gynecologic (if female), ocular, or infectious disease, or signs of acute illness.
* Any medication (including over the counter products and any other herbal/alternative remedies such as St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Screening to Day 28

SECONDARY OUTCOMES:
Assessment of pharmacokinetic (PK) parameter: Cmax | Baseline to 96 hrs
  Maximum plasma concentration
Assessment of PK parameter: AUC | Baseline to 96 hrs
  Area under the plasma concentration versus time curve (AUC)
Assessment of PK parameter: tmax | Baseline to 96 hrs
  Time to reach Cmax
Assessment of pharmacodynamics (PD): glucose profile | Baseline to 24 hrs
  Change from baseline in glucose profile
Assessment of PD: insulin profile | Baseline to 24 hrs
  Change from baseline in insulin profile
Assessment of PD: C-peptide profile | Baseline to 24 hrs
  Change from baseline in C-peptide profile

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site number 8400001, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Bossart M, Wagner M, Elvert R, Evers A, Hubschle T, Kloeckener T, Lorenz K, Moessinger C, Eriksson O, Velikyan I, Pierrou S, Johansson L, Dietert G, Dietz-Baum Y, Kissner T, Nowotny I, Einig C, Jan C, Rharbaoui F, Gassenhuber J, Prochnow HP, Agueusop I, Porksen N, Smith WB, Nitsche A, Konkar A. Effects on weight loss and glycemic control with SAR441255, a potent unimolecular peptide GLP-1/GIP/GCG receptor triagonist. Cell Metab. 2022 Jan 4;34(1):59-74.e10. doi: 10.1016/j.cmet.2021.12.005. Epub 2021 Dec 20. PMID 34932984
- See also: TDU15478 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25355&tenant=MT_SNY_9011